CLINICAL TRIAL: NCT05533294
Title: A Phase 1 Study Evaluating the Effects of ARO-RAGE Injection for Subcutaneous Administration in Healthy Subjects
Brief Title: Study of ARO-RAGE in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARORAGE-1002
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-RAGE (Experimental): single or multiple doses of ARO-RAGE by subcutaneous (sc) injection
  Interventions: Drug: ARO-RAGE Injection
- Placebo (Placebo Comparator): placebo calculated volume to match active treatment by sc injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-RAGE Injection — ARO-RAGE injection for sc administration
  Arms: ARO-RAGE
Drug: Placebo — normal saline (0.9% NaCl) by sc injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single- and multiple-ascending doses of ARO-RAGE Injection in normal healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Normal pulmonary function tests at Screening prior to sputum induction
* Normal 12-lead electrocardiogram (ECG) at Screening
* Non-smoking
* Able to produce an induced sputum sample at Screening
* Participants of child-bearing potential (male and female) must use highly effective contraception and cannot donate sperm or eggs during the study or for at least 12 weeks following the end of the study or last dose of study drug, whichever is later. Women must have a negative pregnancy test and cannot be breastfeeding
* Willing to provide written informed consent and to comply with study requirements

Exclusion Criteria:

* Acute lower respiratory infection within 30 days prior to first dose and/or acute upper respiratory infection within 7 days prior to first dose
* Positive COVID-19 test during Screening window
* Chronic or acute infection that is clinically significant or requires treatment with systemic antibiotics, antivirals, antifungals, or antiparasitics within 30 days prior to first dose
* Any history of chronic pulmonary disease
* Use of immunosuppressive medication within 90 days prior to first dose
* Receipt of any intranasal vaccine within 30 days prior to first dose
* Human Immunodeficiency virus (HIV) infection, seropositive fo Hepatitis B Virus (HBV), seropositive for Hepatitis C Virus (HCV)
* Uncontrolled hypertension
* Use of illicit drugs
* Unwilling to limit alcohol consumption to within moderate limits for the duration of the study
* Use of an investigational agent or device within 30 days prior to first dose
* Prior use of any formulation of ARO-RAGE

Note: additional inclusion/exclusion criteria may apply per protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | From first dose of study drug through the end of study (EOS; up to 113 days or until serum soluble receptor for advance glycation end products [SRAGE] is ≥70% of baseline value, whichever is later)

SECONDARY OUTCOMES:
Change from Baseline Over Time in Forced Expiratory Volume (FEV1) | Baseline through EOS (up to 113 days or until serum SRAGE is ≥70% of baseline value, whichever is later)
Change from Baseline Over Time in Forced Vital Capacity (FVC) | Baseline through EOS (up to 113 days or until serum SRAGE is ≥70% of baseline value, whichever is later)
Change from Baseline Over Time in Diffusing Capacity for Carbon Monoxide (DLCO) | Baseline through EOS (up to 113 days or until serum SRAGE is ≥70% of baseline value, whichever is later)
PK of ARO-RAGE: Maximum Observed Plasma Concentration (Cmax) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29
PK of ARO-RAGE: Area Under the Plasma Concentration versus Time Curve From Zero to 24 Hours (AUC0-24) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29
PK of ARO-RAGE: Area Under the Plasma Concentration versus Time Curve From Zero to the Last Quantifiable Plasma Concentration (AUClast) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29
PK of ARO-RAGE: Area Under the Plasma Concentration versus Time Curve From Zero to Infinity (AUCinf) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29
PK of ARO-RAGE: Terminal Elimination Half-Life (t1/2) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29
PK of ARO-RAGE: Apparent Systemic Clearance (CL/F) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29
PK of ARO-RAGE: Apparent Terminal-Phase Volume of Distribution (VZ/F) | single dose phase: up to 48 hours post-dose; multiple dose phase: up to 6 hours post-dose on Days 1 and 15 or 29

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Grafton, Aukland, New Zealand

IPD SHARING:
Plan to Share IPD: No